CLINICAL TRIAL: NCT05469035
Title: Hamidiye Faculty of Nursing, University of Health Sciences
Brief Title: The Effect of Nurse Training on the Improvement of Subcutaneous Heparin Applications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Associate Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1640
Record Dates: First submitted 2022-06-30; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Nursing Care
Keywords: Subcutaneous heparin injections, nursing, training

STUDY DESIGN:
Intervention Model Description: A randomized controlled, pre-post-test, mixed-method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Nurses in the experimental group participated in mobile-based video learning.
  Interventions: Other: Mobile-based video
- Control (Active Comparator): Nurses in the experimental group participated in face-to-face learning.
  Interventions: Other: Face-to-face

INTERVENTIONS:
Other: Mobile-based video — Nurses in the experimental group participated in mobile-based video learning.
  Other Names: SC Heparin Interventions
  Arms: Experimental
Other: Face-to-face — Nurses in the experimental group participated in face-to-face learning.
  Other Names: SC Heparin Interventions
  Arms: Control

SUMMARY:
One of the most important duties and responsibilities of nurses is drug administration. During drug administration, the nurse uses appropriate administration techniques and ensures patient safety by knowing the drugs and their side effects. This study aimed to examine the effect of nurse training on the improvement of subcutaneous heparin applications. In this study, it was planned to train nurses by using two different training methods. These methods are online and face-to-face training.

In both methods, it was planned to evaluate the subcutaneous drug administration knowledge and skill of nurses before and after the training.

DETAILED DESCRIPTION:
Drug administration is a common nursing clinical intervention. The nurse ensures patient safety by using compatible administration techniques and being aware of the side effects of medications. Pharmacological agents such as heparins, vaccines, insulin, hormone drugs, etc., are generally inappropriate with oral, intravenous or intamuscular intake. Thereupon, they have to be administered by means of subcutaneous (SC) injection. Subcutaneous medications are injected into the tissue layer between the skin and the muscle that is called subcutaneous tissue where does not have a rich blood supply. Suitable areas for subcutaneous injction application are the lateral aspect of the upper arms, posterior aspect of the upper arms, anterior surface of the thigh, unders the scapulas and abdomen in the umbilical region. For the reason that abdominal region has an excess subcutaneous fat tissue, enough space for repeated injections and less muscle activity, it is highly preferred for subcutaneous injections. The angle of entry of the needle into the tissue depends on the needle length and the thickness of the subcutaneous tissue mass. A 90-degree angle is used if the subcutaneous tissue thicknes is about 5 cm. However, when it is 2.5 cm the angle of a 45-degree angle is recommended. To check whether the needle tip is in the vein or not during the application causes the needle movement in the tissue that then results in vascular damage, bleeding, ecchymosis and hematoma formation. Airlock technique in subcutaneous inections is recommended as it ensures that the entire drug is delivered to the tissue as well as preventing the escape of the drug.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study

Exclusion Criteria:

* not have administered subcutaneous heparin in the clinical practice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-08-10 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of subcutaneous heparin applications | Through study completion, an average of 1 months
  The primary outcome of this study is the improvement of nurses' subcutaneous heparin applications. The 25-item checklist prepared by the researchers based on the literature includes the application steps of subcutaneous heparin knowledge and skill.

SECONDARY OUTCOMES:
Comparision of two different method | Through study completion, an average of 1 months
  The secondary outcome of this study is the comparison of the two different education methods.The 25-item checklist prepared by the researchers based on the literature includes the application steps of subcutaneous heparin knowledge and skill.

CONTACTS AND LOCATIONS:
Overall Officials: Demet İnangil, Study Chair — Istanbul Sağlık Bilimleri University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hegland PA, Aarlie H, Stromme H, Jamtvedt G. Simulation-based training for nurses: Systematic review and meta-analysis. Nurse Educ Today. 2017 Jul;54:6-20. doi: 10.1016/j.nedt.2017.04.004. Epub 2017 Apr 19. PMID 28456053